CLINICAL TRIAL: NCT04941573
Title: Assessment of Chronic Lung Allograft Dysfunction Using Single-breath & Multi-breath Hyperpolarized Xenon-129 MRI
Status: Terminated | Type: Observational
Why Stopped: Regulatory Compliance
Sponsor: Xemed LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 834759
Record Dates: First submitted 2021-02-04; First posted 2021-06-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Lung Transplant Rejection
Keywords: CLAD; hyperpolarized xenon MRI; lung transplant; xenon-129 MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (4):
- Post-lung transplant patients not diagnosed with CLAD: This group will have a target enrollment of 50 subjects recruited from the lung transplant patients of pulmonologists from Penn and Temple Lung Transplant Team.
  The subjects will undergo hyperpolarized 129-Xenon MRI and conventional proton MR imaging of the lung at 3, 6, 9, 12, 18, and 24 months following the transplant. Additional pulmonary tests and questionnaires will be performed to assess the lung health status of the patients.
  Interventions: Combination Product: Hyperpolarized 129-Xenon (MagniXene) MRI of the lung
- Post-lung transplant patients diagnosed with CLAD: This group will have a target enrollment of 20 subjects recruited from the lung transplant patients of pulmonologists from Penn and Temple Lung Transplant Team, and whom have been recently diagnosed with CLAD.
  The subjects will undergo a single imaging session of hyperpolarized 129-Xenon MRI and conventional proton MR imaging of the lung.
  Interventions: Combination Product: Hyperpolarized 129-Xenon (MagniXene) MRI of the lung
- Non-transplant COPD patients: This group will have a target enrollment of 10 subjects recruited from the pool of advanced stages of COPD visiting patients from Penn and Temple pulmonologists.
  The subjects will undergo two imaging sessions of hyperpolarized 129-Xenon MRI and conventional proton MR imaging of the lung within approximately week to ensure imaging metric reproducibility.
  Interventions: Combination Product: Hyperpolarized 129-Xenon (MagniXene) MRI of the lung
- Healthy control subjects: This group will have a target enrollment of 10 subjects recruited from general population and not suffering from any chronic lung diseases.
  The subjects will undergo two imaging sessions of hyperpolarized 129-Xenon MRI and conventional proton MR imaging of the lung within approximately week to ensure imaging metric reproducibility.
  Interventions: Combination Product: Hyperpolarized 129-Xenon (MagniXene) MRI of the lung

INTERVENTIONS:
Combination Product: Hyperpolarized 129-Xenon (MagniXene) MRI of the lung — Hyperpolarized xenon is a contrast imaging agent for lung MR imaging. Inert noble gas xenon is hyperpolarized using Xemed developed technology. The gas is administered to the human subjects as a short seconds-long breath-hold while inside the MRI scanner. Once the gas is inhaled, lung images of HP Xenon distributed within the lung spaces can be acquired. Additionally, xenon follows a similar path to oxygen, dissolving in lung tissue and further in bloodstream.

SUMMARY:
This study will use Magnetic Resonance Imaging (MRI) to study the lungs of 90 volunteers using the inhaled contrast agent, hyperpolarized xenon-129. Once inhaled, this gas can provide information to imagers regarding lung functionality across specific regions of the lungs by assessing the replacement of air during the normal breathing cycle, how much oxygen is in the airspaces, and if the natural spongy tissue structure has been compromised by lung disease. Of the 90 subjects, 70 will be patients who received lung transplantation from the Penn/Temple Lung Transplant Teams and are receiving follow up treatment at HUP or TUH, 10 will be healthy control subjects who participated favorably in our HP 129Xe imaging protocol, and 10 will be patients who have been diagnosed with chronic obstructive pulmonary disease (COPD)-preferentially recruited from the Temple University COPDGene cohort, who have never undergone a lung transplant. 20 of the lung transplant recipient subjects will be patients who have received a recent clinical diagnosis of chronic lung allograft dysfunction (CLAD) prior to enrollment in our study, while the other 50 will have recently undergone their initial transplant surgery at the time of enrollment.

DETAILED DESCRIPTION:
This study assesses the operating characteristics of HP 129Xe MRI in an effort to evaluate its performance in identifying early signs of CLAD or graft acceptance in 70 total lung transplant recipients, 20 of whom have been recently diagnosed with CLAD, 10 non-transplant COPD subjects, and 10 healthy control patients. These subjects will be recruited from the patients of transplant pulmonologists on the Penn and Temple Lung Transplant Team. Subjects will be recruited regardless of race or gender. Study visits will last 1-2 hours for each subject and will occur at various time points following their operation. The baseline visit will occur at the conclusion of their 3 month post-transplant visit, with study follow-up visits occurring at the conclusion of the 6, 9, 12, 18, and 24 month post-transplant visit. For the convenience of the subjects, most study visits will begin at the conclusion of their follow-up visit with their transplant pulmonologist. If this does not work for the subject, an alternative date will be scheduled and the PFT's/Physical exam results from the most recent visit with their transplant pulmonologist will be used for that study visit. There will be a 45-day imaging window for each post-transplant visit, allowing MR imaging to be performed within 45 days before or after the anticipated imaging date, granting more flexibility for both subjects and researchers to ensure that each imaging session is successfully completed. If patients decide to not participate in this study, their decision will not affect their standing with HUP or their physician. Both healthy control subjects and non-transplant COPD subjects will be imaged twice within approximately one week to ensure imaging metric reproducibility in both cohorts. Diagnosed CLAD subjects will undergo a single imaging session each. The images of the diagnosed CLAD subjects will serve as a necessary reference for predicting the early decline of lung function in pre-CLAD transplant recipients.

ELIGIBILITY:
General Inclusion Criteria:

* For transplant recipients: the subject is a lung transplant recipient who is over 18 years of age, underwent lung transplantation at the Hospital of the University of Pennsylvania or Temple University Hospital, and is receiving follow up care from the Penn or Temple Lung Transplantation teams following said transplant. Written informed consent will be obtained and documented after the subject receives oral and written information about the study.
* For diagnosed CLAD patients: the subject is a lung transplant recipient who is over 18 years of age, underwent lung transplantation at the Hospital of the University of Pennsylvania or Temple University Hospital, and has recently received a clinical diagnosis of CLAD. Written informed consent will be obtained and documented after the subject receives oral and written information about the study.
* For non-transplant COPD patients: the subject is over 18 years old, has been diagnosed with chronic obstructive pulmonary disease, and has never received a lung transplant.
* For healthy controls: the subject is over 18 years of age.

Exclusion Criteria:

* Patients less than 18 years old
* Patients known to be pregnant - a positive pregnancy test will be used to respectively exclude pregnant patients,
* Any known contraindication to MRI examination
* Anyone with an implanted metal device
* Inability to provide informed consent
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed participation in the study.
* History of uncompensated organ failure (i.e. organ failure that is not stabilized through medical intervention), which will be assessed by the PI.
* Homelessness or other unstable living situation
* Active drug or alcohol dependence
* Claustrophobia
* Subjects weighting more than 300 pounds.
* Subjects with chest size larger than the bore of MRI machine from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients 18-80 years with recent lung transplant diagnosed and not diagnosed with CLAD.
  * Patients 18-80 years with COPD.
  * Healthy subjects 18-80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Number and extent of functional and microstructural abnormalities observed with hyperpolarized xenon-129 in the lung transplant patients. | up to two years after the lung transplant (imaging at 3, 6, 9, 12, 18, and 24 months post-transplant)
  The primary endpoint is the number and extent of functional and microstructural abnormalities observed in the lung transplant recipients following inhalation of polarized 129Xe. For the single-breath protocol, images will be obtained immediately after inhalation and during the subsequent breath hold. During the multi-breath protocol, images will be obtained during a <1 second breath hold at the end of the exhalation. Fractional ventilation will be obtained based on the signal build up for multi-breath breathing of HP 129Xe over the course of the inhalations. Regional alveolar tension of oxygen (PAO2) will be obtained based on the signal decay over time during the breath-hold. ADC will be determined using diffusion sensitizing gradients according to standard imaging protocols. Dissolved phase HP 129Xe will also be obtained by imaging the gas at its different frequencies when bound to hemoglobin and when crossing alveolar walls.

SECONDARY OUTCOMES:
Examine correlations between pulmonary function test scores, questionnaires, and overall scores for the metrics of HP 129Xe MRI ventilation images, ADC, gas exchange, and dissolved phase information. | end of the project data analysis
  The relationship between pulmonary function test scores, overall scores of the ventilation images, ADC gas exchange scores, and dissolved phase information generated during HP 129Xe MR imaging will be examined. The statistical plan for the secondary study endpoints will be to use a simple two-sided t-test to see if there are detectable differences between our values within the same patient and their MRI values between the two gases. In this case, the t-test is paired, as we are looking at variables in the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Itkin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States